CLINICAL TRIAL: NCT06149247
Title: Pilot Study of HyBryte (Synthetic Hypericin) Versus Valchlor (Mechlorethamine) in the Treatment of CTCL
Brief Title: HyBryte (Synthetic Hypericin) Versus Valchlor (Mechlorethamine) in the Treatment of CTCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soligenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPN-CTCL-04
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Cutaneous T-Cell Lymphoma/Mycosis Fungoides
Keywords: CTCL; MF; Hypericin; HyBryte
MeSH Terms: conditions — Mycosis Fungoides | interventions — hypericin; Amines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HyBryte (0.25 % hypericin) (Experimental): HyBryte (0.25 % hypericin) ointment will be applied to CTCL lesions and treated with visible light 18-24 hours later starting at 6 J/cm^2. Drug application/light session will be done twice a week (at least 2 calendar days apart) for 12 weeks.
  Interventions: Drug: Hypericin
- Valchlor (mechlorethamine) (Active Comparator): Valchlor (0.016% mechlorethamine) gel will be applied to CTCL lesions once daily for 12 weeks.
  Interventions: Drug: Mechlorethamine Topical Gel

INTERVENTIONS:
Drug: Hypericin — HyBryte is synthetic hypericin formulated as a 0.25% hypericin ointment.
  Other Names: HyBryte; SGX301
  Arms: HyBryte (0.25 % hypericin)
Drug: Mechlorethamine Topical Gel — Valchlor is an FDA-approved drug for the treatment of CTCL.
  Other Names: Valchlor
  Arms: Valchlor (mechlorethamine)

SUMMARY:
The objective of this clinical study is to compare the safety and effectiveness of Valchlor versus HyBryte following 12 weeks of treatment.

DETAILED DESCRIPTION:
Participants will be randomized to receive HyBryte or Valchlor in a 1:1 randomization. Participants will be treated for 12 weeks and follow-up visits will be conducted 1, 2, and 4 weeks after completion of the treatment phase of the trial.

Prior to randomization, each participant will have at least 3 and up to 5 lesions identified (index lesions) that will be evaluated during the treatment phase and during the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 3 active treatment-accessible CTCL lesions
* Subjects must have a clinical diagnosis of cutaneous T-cell lymphoma (CTCL, mycosis fungoides), Stage IA, IB, or Stage IIA
* Subjects willing to follow the clinical protocol and voluntarily give their written informed consent
* Female subjects not pregnant nor nursing and willing to undergo a pregnancy test within 30 days prior to treatment initiation

Exclusion Criteria:

* History of severe allergic reaction to any of the components of HyBryte or mechlorethamine (Valchlor)
* Pregnancy or mothers who are breast-feeding
* All women of childbearing potential (WOCBP) and males with female partners who are WOCBP not willing to use effective contraception
* Subjects with history of sun hypersensitivity or photosensitive dermatoses (eg, porphyria, systemic lupus erythematosus (SLE), Sjogren's syndrome, etc.)
* Subjects whose condition is spontaneously improving
* Subjects receiving Valchlor (or any topical compound containing Mechlorethamine) in the preceding 2 months
* Subjects receiving topical steroids or other topical treatments (eg, targretin gel) on treatment accessible lesions for CTCL within 2 weeks of enrollment
* Subjects receiving systemic steroids, psoralen ultraviolet A (UVA) radiation therapy (PUVA), narrow band ultraviolet B (UVB) light therapy (NB-UVB) or carmustine (BCNU) or other systemic therapies for CTCL within 3 weeks of enrollment
* Subjects who have received electron beam irradiation within 3 months of enrollment
* Subjects with a history of significant systemic immunosuppression
* Subjects taking other investigational drugs or drugs of abuse within 30 days of enrollment
* Subject has any condition that, in the judgment of the Investigator, is likely to interfere with participation in the study
* Subjects receiving drugs known to cause photosensitization within 2 weeks of starting HyBryte therapy unless they have not had evidence of photosensitization after receiving a stable dose of the medication for a minimum of 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester Skin Lymphoma Medical Group, Fairport, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HyBryte (0.25 % Hypericin) | Valchlor (Mechlorethamine)
Started | 5 | 5
Completed | 5 | 4
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HyBryte (0.25 % Hypericin) | Valchlor (Mechlorethamine) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (19.18) | 62.4 (13.48) | 59.3 (16.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Treatment Response in the Modified Composite Assessment of Index Lesion Disease Severity (mCAILS) Score
Description: A treatment response is defined as a ≥50% improvement in mCAILS score at Week 12 when compared to the mCAILS score at baseline.
  The Modified Composite Assessment of Index Lesion Disease Severity (mCAILS) score measures: Erythema (or redness) on a scale of 0 (no redness) to 8 (very red), Scaling on a scale of 0 (no scaling) to 8 (all of the lesion is covered by a very rough surface), Plaque Elevation on a scale of 0 (no evidence of plaque above normal skin level) to 3 (plaque shows marked elevation above normal skin level) and Surface Area on a scale of 0 (no lesion/surface area is 0 cm^2) to 18 (the lesion is larger than 300 cm^2). A lower score means a better outcome.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HyBryte (0.25 % Hypericin) | Valchlor (Mechlorethamine)
Number analyzed (Participants) | 5 | 5
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 16 weeks
Arm/Group | HyBryte (0.25 % Hypericin) | Valchlor (Mechlorethamine)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HyBryte (0.25 % Hypericin) (N=5) | Valchlor (Mechlorethamine) (N=5)
Swollen lymph nodes (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Allergic contact dermatitis (General disorders) | 0 (0) | 1 (1)
Dermatitis (General disorders) | 0 (0) | 1 (1)
Rash (General disorders) | 0 (0) | 1 (1)
Sensitivity (General disorders) | 0 (0) | 1 (1)
COVID-19 infection (Infections and infestations) | 1 (1) | 0 (0)
Neck pain/inflammation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Id reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT06149247/Prot_SAP_000.pdf